CLINICAL TRIAL: NCT03730519
Title: Investigation of the Efficacy and Safety of Baroreflex Activation Therapy in Patients With Refractory Hypertension and Those With Highly Variable Blood Pressure Due to Peripheral Baroreflex Failure
Brief Title: UK Registry for Baroreflex Activation Therapy
Acronym: UK-BAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the pandemic
Sponsor: Queen Mary University of London (Other)
Collaborators: CVRx, Inc. (Industry)
Responsible Party: Principal Investigator, Melvin D Lobo, Professor, Queen Mary University of London
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCPG1M8R
Record Dates: First submitted 2018-10-16; First posted 2018-11-05 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Baroreflex Failure Syndrome; Hypertension, Resistant to Conventional Therapy
Keywords: Refractory Hypertension
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Hypertension

STUDY DESIGN:
Intervention Model Description: This study is a post-marketing open label twin arm, single centre clinical trial of electrical carotid sinus stimulation with the Barostim Neo device to target sub-optimally controlled arterial hypertension or highly variable blood pressure in patients for whom no alternative therapies are available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with refractory hypertension (Active Comparator): Patients with refractory hypertension which cannot be controlled with drug therapy in the hands of hypertension specialists will be treated with Baroreflex Activation Therapy with Barostim Neo and followed up for a period of up to 3 years
  Interventions: Device: Baroreflex Activation Therapy with Barostim Neo
- Patients with highly variable BP (Active Comparator): Patients with symptomatic highly variable blood pressure due to afferent baroreceptor failure which cannot be controlled with drug therapy in the hands of hypertension specialists will be treated with Baroreflex Activation Therapy with Barostim Neo and followed up for a period of up to 3 years
  Interventions: Device: Baroreflex Activation Therapy with Barostim Neo

INTERVENTIONS:
Device: Baroreflex Activation Therapy with Barostim Neo — Baroreflex activation therapy (BAT) delivers electrical field stimulation at the carotid sinus to lower BP.
  Other Names: Electrical Carotid sinus stimulation

SUMMARY:
This study is a post-marketing open label single arm, single centre clinical trial of electrical carotid sinus stimulation with the Barostim Neo device to target sub-optimally controlled arterial hypertension or highly variable blood pressure in patients for whom no alternative therapies are available.

DETAILED DESCRIPTION:
Hypertension is a major health issue globally and is the number one risk factor for cardiovascular morbidity and mortality. Despite decades of innovation in pharmacotherapeutics, suboptimal BP control remains a problem worldwide. Alternative therapies for hypertension are therefore urgently needed.

This project addresses the following important unmet needs:

1. . Refractory hypertension may respond to device based approaches such as baroreflex activation therapy (BAT) but further independent research is needed to clarify the role of novel technologies. It is not possible to undertake research into BAT at all due to lack of funding and the manufacturer is not undertaking clinical trials of the therapy in the UK.
2. . Patients with highly variable BP disorders constitute a very small but important sub-group of the hypertensive population but are the most challenging to manage as no drug therapy exists to combat high and low BP simultaneously. This group of patients have very poor quality of life and are unable to work due to their profound BP variability. Many of them experience frequent hospital admissions for lengthy periods as a result of potentially life-threatening hypertension. Treatment with BAT may feasibly improve management of their condition by dampening BP variability and preventing hypertensive surges whilst allowing the patients to continue with measures to prevent hypotension using compression hosiery and drugs.

This project has the following objectives

Primary:

To establish a UK national registry for treatment of blood pressure disorders with baroreflex activation therapy in the following patient groups:

* Patients with refractory hypertension (Ref-HTN) regardless of pharmacotherapy (up to 15 patients)
* Patients with highly variable BP disorders (BPV) the aetiology of which indicates that peripheral baroreflex failure is the underlying diagnosis (up to 10 patients)

Secondary

* To undertake mechanistic research to better understand the mechanism of action of baroreflex activation therapy and the role of the baroreflex in hypertensive disorders by measuring indices of autonomic function (parasympathetic and sympathetic nervous system tone) and humoral factors such as renin/aldosterone and copeptin in response to BAT.
* To position the Barts BP Clinic as a national referral centre for the management of complex circulatory disorders with access to experimental treatments unavailable elsewhere in the UK.
* To foster a more 'joined up' approach to BAT by promoting awareness of its benefits among primary care practitioners and other secondary care specialists.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be enrolled following an informed consent. The subject will be able to understand and comply with protocol requirements, instructions and protocol restrictions.
2. The study subjects will be either:

   I. Refractory hypertensive patients (daytime systolic ambulatory BP (ABP) > 150 mmHg) in whom all pharmacological approaches to control BP have failed or were intolerable.

   or II. Symptomatic patients with exaggerated BPV documented on daytime ABP monitoring (SD >18 mmHg) who cannot achieve effective BP control with pharmacological approaches
3. For BPV group, evidence of peripheral baroreflex dysfunction as determined by non-invasive autonomic function testing
4. Patients will have been established on a stable antihypertensive treatment regime for at least 1 month by the time of participation in the study and changes in pharmacological intervention for the duration of the trial are to be avoided unless clinically mandated.

Exclusion Criteria:

* HTN secondary to an identifiable and treatable cause
* Carotid atherosclerosis determined by ultrasound or angiographic evaluation greater than 50% stenosis
* Ulcerative plaques in the carotid artery as determined by ultrasound or angiographic evaluation
* Bifurcation of the carotid on the side planned needs to be below level of mandible by ultrasound
* Uncontrolled, symptomatic cardiac bradyarrhythmias.
* Myocardial infarction, unstable angina or cerebral vascular accident within 3 months before implant.
* Clinically significant cardiac valvular disease
* Prior implant in the carotid sinus region,
* Currently implanted electrical medical devices,
* End stage renal (with eGFR <15 mL/min) or liver disease
* Pregnancy or contemplating pregnancy.
* BMI > 40 kg/sq m
* Inability to tolerate ambulatory blood pressure monitoring
* Patient with other co-morbidity likely to have life expectancy <3y
* Systolic left heart failure with ejection fraction <40%

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Ambulatory Systolic & Diastolic Blood Pressure changes in patients with uncontrolled (refractory) hypertension | 6 months
Ambulatory Systolic & Diastolic Blood Pressure variability change in patients with highly variable BP due to baroreflex failure | 6 months
Incidence of Treatment-Emergent Adverse Events in both groups of patients | 6 months

SECONDARY OUTCOMES:
Change in European Quality of Life 5 dimension (Eq-5D) score in both groups of patients | 6 months
  Eq5D is a standardised/validated instrument to assess health outcome. It consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a self-rated health scale on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. An Eq5D index of 1.0 indicates full health, and -0.59 denoted death
Changes in autonomic indices in both groups of patients | 6 months
  Non-invasive measurement of parasympathetic (vagal) tone and sympathetic tone using a Neuroscope measurement device with real time beat to beat BP measurement

OTHER OUTCOMES:
Change in echocardiographic left ventricular mass in both groups of patients | 6 months
Change in pulse wave velocity in both groups of patients | 6 months
Change in antihypertensive whole medicine equivalent in both groups of patients | 6 months
  For each patient, the sum of the percentage of the maximum licensed dose (MLD) for each medicine gives the total whole medicine equivalent (WME).

CONTACTS AND LOCATIONS:
Overall Officials: Melvin D Lobo, MBChB PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- William Harvey Research Institute, London, United Kingdom